CLINICAL TRIAL: NCT00264108
Title: EPREX (Epoetin Alfa) Versus ARANESP (Darbepoetin Alfa): Looking at Outcome of Anemia Treatment and Comparing Cost-effectiveness (EVALUATE).
Brief Title: Cost-effectiveness Study of Epoetin Alfa and Darbepoetin Alfa in Adult Patients With Cancer Who Have Anemia
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag B.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR002455; EPOCAN4015
Record Dates: First submitted 2005-12-09; First posted 2005-12-12 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Anemia; Neoplasms
Keywords: Antineoplastic agents; Chemotherapy; Cost-effectiveness; Epoetin alfa; Darbepoetin alfa
MeSH Terms: conditions — Anemia; Neoplasms | interventions — Darbepoetin alfa; Epoetin Alfa

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: Epoetin alfa 40 000 IU once weekly variable treatment length.
  Interventions: Drug: Epoetin alfa
- 2: Darbepoetin alfa Either 150 ug once weekly or 500 ug once every 3 wks variable treatment length.
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Darbepoetin alfa — Either 150 ug once weekly or 500 ug once every 3 wks, variable treatment length.
  Groups: 2
Drug: Epoetin alfa — 40,000 IU once weekly, variable treatment length.
  Groups: 1

SUMMARY:
The purpose of this study is to evaluate the cost-effectiveness of epoetin alfa compared with darbepoetin alfa in the treatment of anemia in adults receiving chemotherapy for cancer. Epoetin alfa and darbepoetin alfa are genetically engineered proteins that stimulate red blood cell production.

DETAILED DESCRIPTION:
Anemia has been identified as a common complication and a widespread problem in the cancer population. Anemia is a condition in which a patient has below normal levels of hemoglobin, the substance in red blood cells that carries oxygen to all parts of the body. People with severe anemia may experience fatigue and shortness of breath with activity. Therefore, this condition can have a negative influence on a person's quality of life. Epoetin alfa and darbepoetin alfa, used to treat anemia in cancer patients, are genetically engineered proteins that stimulate red blood cell production. This study investigates treatment of anemia using either epoetin alfa or darbepoetin alfa during chemotherapy in adult patients with cancer. The study is intended to collect information on normal medical practice and routine anemia management performed at the participating centers. This is an observational, non-randomized, prospective, comparative, parallel-group survey performed in The Netherlands. Patients with various severities of disease may enter the survey as soon as either their epoetin alfa or their darbepoetin alfa treatment starts and will be followed until the end of their epoetin alfa/darbepoetin alfa treatment. Patient data are collected, on average, once monthly (depending on the treatment being received) and this continues until 4 weeks after the end of treatment with epoetin alfa or darbepoetin alfa. An assessment of cost-effectiveness will be made for both treatments. The assessment of cost-effectiveness will be based on the following: cancer type and status, chemotherapy and other anti-cancer treatment, hemoglobin levels, use of either epoetin alfa or darbepoetin alfa, use of blood transfusions, and serum iron levels and iron supplementation. Safety evaluations include the incidence of serious and non-serious adverse events. Because the study involves only collection of information, no treatment will be required by the Sponsor and no medication will be supplied by the Sponsor. Epoetin alpha and darbepoetin alpha are administered according to routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of solid tumors, multiple myeloma (Kahlers' disease), non-Hodgkin lymphoma or Hodgkins' disease
* Patients must already be receiving chemotherapy or start their first cycle within a week of enrollment
* Patients must receive either epoetin alfa or darbepoetin alfa treatment (expected treatment duration is at least 4 weeks)

Exclusion Criteria:

* Patients not meeting all of the inclusion criteria for entry into the study
* Patients who cannot read the Dutch language and/or do not understand the Dutch Informed Consent Form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients receiving epoetin- or darbepoetin alfa as anemia treatment during chemotherapy, as part of the common practice of participating physicians. Patients may enter the study as soon as either their epoetin alfa or their darbepoetin alfa treatment starts.
Sampling Method: Non-Probability Sample
Enrollment: 492 (Actual)
Dates: Start 2005-06; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Cost-effectiveness based on: cancer type and status, chemotherapy and other anti-cancer treatment, hemoglobin levels, use of either epoetin alfa or darbepoetin alfa, use of blood transfusions, serum iron levels and iron supplementation. | 4 weeks, 8 weeks and end of treatment

SECONDARY OUTCOMES:
Safety evaluations including the incidence of serious and non-serious adverse events. | from start of (Darb)epoetin treatment to end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag B.V. Clinical Trial, Study Director — Janssen-Cilag B.V.
Locations (20):
- Netherlands (20):
  - 's-Hertogenbosch
  - Amstelveen
  - Amsterdam
  - Bergen op Zoom
  - Den Helder
  - Dirksland
  - Ede Gld
  - Eindhoven
  - Goes
  - Gorinchem
  - Helmond
  - Hoofddorp
  - Meppel
  - Purmerend
  - Rotterdam
  - Spijkenisse
  - Tilburg
  - Utrecht
  - Winterswijk
  - Zeist